CLINICAL TRIAL: NCT02445482
Title: SOLTI Molecular Screening Program: a Pilot Study to Implement Personalized Therapy for Patients With Advanced or Metastatic Breast Cancer
Brief Title: SOLTI Breast Cancer Molecular Screening Program (AGATA)
Acronym: AGATA
Status: Completed | Type: Observational
Sponsor: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: SOLTI-1301
Record Dates: First submitted 2015-01-13; First posted 2015-05-15 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of the archived initial or metastatic tumor sample (one 60 μm formalin-fixed, paraffin-embedded tumor block). If archived material is not available, a biopsy of the metastatic cancer should be performed to obtain such material
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Biopsy — archival tissue or fresh biospsy

SUMMARY:
In recent years, the advance in high-throughput techniques, such as microarrays and next gen sequencing (NGS) technologies, have allowed a more precise classification of the breast cancer molecular subtypes and a more personalized approach to anti-cancer therapy. To date, conventional methods to select patients for clinical trials with anti-targeted agents according to molecular criteria are generally limited to the analysis of a few biomarkers. Recent studies have shown how this strategy is inappropriate in case of infrequent molecular alterations and that the ideal strategy would consist in simultaneous examination of large numbers of actionable genomic alterations.

This is the first genomic screening platform ever attempted in Spain. By this molecular platform SOLTI aims to increase the likelihood of a patient being included in a trial designed specifically for her molecular tumor type. Thus, the primary objective of this pilot study is to determine the Platform's effectiveness to include patients in clinical trials with targeted agents based on the tumor molecular profiling.

DETAILED DESCRIPTION:
This is a prospective, multicenter, pilot study conducted in eight sites located in Spain. Up to 260 female or male patients, between 18-70 years with advanced or metastatic breast cancer will be screened. These patients will be about to receive, or receiving, or will have received treatment for their disease in either a clinical trial or the healthcare setting. Quality of life score according to ECOG scale ≤ 2 and a minimal life expectancy of 3 months. Upon signed inform consent and confirmation of eligibility criteria, tumor samples will be obtained from the patients either by biopsy of metastatic cancer or from archived tissue previously available at the site, and their genomic profile will be analyzed. It will be assessed the mutational status of a panel of genes considered relevant to the tumor biology and treatment. Detected variants /mutations in samples will not be classified according to their origin somatic or germline, since no normal paired DNA will be analyzed. Should any clinical trial match the patient's molecular profile, she/he will be offered to participate in it and the available samples left after sequencing will be supplied when a central confirmation would be requested. The patient's clinical data will be collected on a quarterly basis until death or consent withdrawal.

Mutation testing will be carried out at three laboratories experienced in high-throughput sequencing techniques: the VHIO Cancer Genomics Core laboratory of Barcelona, at Genomics Laboratory of the Research Institute of the Doce de Octubre University Hospital of Madrid and at the Genomics laboratory of the University Clinical Hospital of Valencia. There is a need to join efforts, set standards and optimize procedures for the benefit of all patients, so that the opportunity to participate in a genomic screening program can be offered to the great majority of hospitals that lack the technology required for these tests.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male patients
* Between 18 and 70 years of age
* Signed informed consent prior to any screening procedure
* Advanced or Metastatic breast cancer of any subtype confirmed both pathologically and radiologically (stage IIIb- IV disease)
* The patient may present with a responding, stable or progressive disease
* The subjects must be about to receive, or receiving, or will have completed treatment for their metastatic disease with any line of treatment in either a clinical trial or the healthcare setting
* Availability of one archived initial or metastatic tumor sample. If archived material were not available, a biopsy of the metastatic cancer should be performed to obtain such material.
* Measurable or non-measurable disease
* Quality of life score according to ECOG scale ≤ 2
* Minimal life expectancy of 3 months

Exclusion Criteria:

* Presence of progressive disease at the time of inclusion requiring treatment initiation before genomic profile results are obtained
* LVEF<50% (MUGA)
* Inadequate bone marrow reserve or organ dysfunction shown by any of the following laboratory values:
* Absolute neutrophil count
* Platelet count< 100 x 109/L
* Hemoglobin < 90 g/dL
* AST/ALT > 2.5 times the upper limit of normality if no demonstrable hepatic metastases, or > 5 times the upper limit of normality in the presence of hepatic metastases
* Total bilirubin > 1.5 times the upper limit of normality
* Creatinine>1.5 times the upper limit of normal
* Corrected calcium > upper limit of normality
* Phosphate > upper limit of normality
* Presence of any other type of cancer, except suitably

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in eight sites located in Spain, and up to 260 patients with advanced or metastatic breast cancer will be screened. These patients will be about to receive, or receiving, or will have received treatment for their disease in either a clinical trial or the healthcare setting
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Platform's effectiveness mesured as the proportion of patients included in clinical trials with targeted agents based on the tumor molecular profiling | 30 months

SECONDARY OUTCOMES:
Characterization of the genomic profiles of the breast cancer patients included in the program listing the percentage of mutations deemed potentially actionable | 30 months
List of the potential barriers of the program | 30 months
Comparison of the percentage of patients included in clinical trials according to their genomic profile between the different panels and sequencing methods. | 30 months
Percentage of the patients alive and without progression (PFS) and percentage of patients alive (OS) of the patients receiving any targeted therapy based on molecular profiling | 30 months
Comparison of the PFS and OS percentages of patients included in clinical trials according to the genomic profile of their tumor with those of patients not assigned to these clinical trials | 30 motnhs

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ciruelos, MD, Principal Investigator — SOLTI Breast Cancer Research Group; Sonia Pernas, MD, Principal Investigator — SOLTI Breast Cancer Research Group
Locations (10):
- Spain (10):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Català d' Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Vall d' Hebrón, Barcelona
  - Institut Català d' Oncologia de Girona, Girona
  - Complejo Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hoapital Universitario Arnau de Vilanova, Valencia
  - Hospital Universitario Clinic de Valencia, Valencia